CLINICAL TRIAL: NCT03272074
Title: Egg Consumption Positively Affects Glycemic Control and Insulin Sensitivity in Individuals With Pre- and Type II-diabetes
Brief Title: Egg Consumption and Glycemic Control in Individuals With Pre- and Type II-diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Egg Nutrition Center (Other)
Responsible Party: Principal Investigator, Bahram Arjmandi, Margaret A. Sitton Professor, Director of Center for Advancing Exercise and Nutrition Research on Aging, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015.15638
Record Dates: First submitted 2017-08-28; First posted 2017-09-05 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus, Type 2; Obesity; Pre Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Glucose Intolerance | interventions — Egg White

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Egg Group (Group A) (Experimental): Participants will consume one large egg per day for 12 weeks
  Interventions: Other: Egg and egg white
- Egg White Group (Group B) (Active Comparator): Participants will consume equivalent amounts of egg whites for 12 weeks
  Interventions: Other: Egg and egg white

INTERVENTIONS:
Other: Egg and egg white — Participants will consume either one large eggs or equivalent amount of egg white (3/4 cups) for 12 weeks. Participants will maintain their regular diet and physical activities.

SUMMARY:
The intent of this study is to examine the extent to which daily incorporation of egg into a diet improves glycemic control, insulin sensitivity, lipid profiles, and body composition in overweight and obese adults with pre- and type II-diabetes. The hypothesis of this study is that the daily incorporation of one large egg into a diet for 12 weeks will exert positive effects on factors associated with glycemic control and insulin sensitivity in overweight and obese adults with pre- and type II-diabetes through improvements in body weight, body composition, and lipid metabolism.

DETAILED DESCRIPTION:
Pre-diabetes is a condition that is characterized by elevated fasting blood glucose levels secondary to insulin resistance; however, fasting blood glucose levels are not elevated to the extent where it can be classified as type II-diabetes. Pre-diabetes may lead to type II-diabetes and is estimated to do so at an annual rate of approximately 10% in the United States (US) where approximately 79 million individuals have been diagnosed with pre-diabetes. In addition, most of the individuals presenting with pre-diabetes are overweight or obese, which makes long-term weight management an essential component in reducing the development of diabetes. Eggs are a rich source of important nutrients such as vitamins, minerals, proteins, carotenoids, choline, and lecithin. Many of the nutrients found in eggs function as antioxidants or as an essential component of antioxidants. Several studies have demonstrated that the onset and progression of diabetes are associated with increased oxidative stress. In vitro studies have shown that high-density lipoprotein (HDL) acts as a buffer mechanism for oxidative stress and inflammation due to its antioxidant effects. Thus, high blood levels of HDL may reduce insulin resistance and subsequently the development of type II-diabetes through its antioxidant and anti-inflammatory effects. Additionally, HDL can exert beneficial effects on glucose levels through the apolipoprotein A-1 (Apo A) action which increases glucose uptake by increasing insulin secretion in pancreatic beta cells. Because the development of diabetes involves an interaction between genetic predisposition and environmental factors including and excessive body weight, and eggs have been shown to positively influence body composition, we believe that eggs can improve glycemic control, insulin sensitivity, and lipid profiles through improvements in weight and body composition. To our knowledge, there have not been any studies investigating the effects of dietary egg consumption on improving glycemic control, insulin sensitivity, lipid profiles, and body composition in overweight and obese adults with pre- and type II-diabetics. Our long-term goal is to bring forth evidence that the regular consumption of eggs is effective in reducing insulin resistance and subsequently the incidence of pre-diabetes and type II-diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Overweight and obese, BMI is between 25 kg/m2 and 45 kg/m2
* With pre- and type II-diabetes. Subjects will be eligible if their Hgb A1c level is >5.6%

Exclusion Criteria:

* Subjects with BMI≤ 24 or ≥46 kg/m2
* Uncontrolled hypertension (≥160/100 mmHg), active cancer, asthma, thyroid, glaucoma, kidney, liver and pancreatic diseases will be excluded from the study.
* Subjects who are participating in any weight loss program and/or are heavy smokers (more than 20 cigarettes per day) will be excluded from the study.
* Subjects who are allergic to egg and egg products will also be excluded from the study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-09-11 (Actual); Primary Completion 2016-09-07 (Actual); Study Completion 2017-08-05 (Actual)

PRIMARY OUTCOMES:
Fasting blood glucose, insulin resistance, and insulin sensitivity | 12 weeks
  Commercially available enzyme-linked immunosorbent assay (ELISA) kits will be used to measure fasting blood glucose levels (mg/dL.). Insulin levels will be measured using a commercially available ELISA kit (mg/dL). blood glucose and insulin level measurements will be used to calculate Insulin sensitivity and insulin resistance will be measured using HOMA-IR and HOMA-β using the HOMA2 Calculator v2.2.2

SECONDARY OUTCOMES:
Lipid panel | 12 weeks
  ELISA kits will be used to measure the lipid panel parameters (mg/dL)

OTHER OUTCOMES:
Body composition | 12 weeks
  A certified operator will obtain DXA scans of each subject using DXA (GE Healthcare Lunar, Madison, WI, U.S.).
ABCA1 Protein | 12 weeks
  ELISA kits will be used to measure the ABCA1 protein (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Shirin Pourafshar, PhD, Study Director — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No